CLINICAL TRIAL: NCT04760730
Title: A Phase I/II Single-Blinded Randomised Safety and Immunogenicity Study in Adults of AZD1222 and rAd26-S Administered as Heterologous Prime Boost Regimen for the Prevention of COVID-19
Brief Title: Safety and Immunogenicity Study in Adults of AZD1222 and rAd26-S Administered as Heterologous Prime Boost Regimen for the Prevention of Coronavirus Disease 2019 (COVID-19)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CV03872091
Record Dates: First submitted 2021-02-17; First posted 2021-02-18 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Severe acute respiratory syndrome coronavirus 2; 2019-nCoV; 2019 novel coronavirus; Respiratory disease; lung disease; COVID-19 Pandemic; coronavirus
MeSH Terms: conditions — COVID-19; Respiration Disorders; Lung Diseases; Coronavirus Infections | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Who Masked: Participant
Masking Description: single-blinded (participant-blinded study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: 1 intramuscular (IM) injection of AZD1222 on Day 1 followed by rAd26-S on Day 29 (Experimental): Subjects will receive 1 intramuscular (IM) injection of 5 × 10^10 viral particles (vp) (nominal) of AZD1222 on Day 1 followed by rAd26-S (1.0±0.5) х 10^11 viral particles (vp) (nominal) on Day 29
  Interventions: Biological: AZD1222; Biological: rAd26-S
- Group B: 1 intramuscular (IM) injection of rAd26-S on Day 1 followed by AZD1222 on Day 29 (Experimental): Subjects will receive 1 intramuscular (IM) injection of rAd26-S (1.0±0.5) х 10^11 viral particles (vp) (nominal) on Day 1 followed by AZD1222 5 × 10^10 vp (nominal) on Day 29.
  Interventions: Biological: AZD1222; Biological: rAd26-S

INTERVENTIONS:
Biological: AZD1222 — Active substance: ChAdOx1 nCoV-19, a replicant-deficient simian adenoviral vector in the amount of 5 х 10^10 particles (nominal) per dose (unit dose strength > 0.7 × 10^11 vp/mL).
  Solution for intramuscular injection, supplied in vials in a carton box
  Other Names: ChAdOx1 nCoV-19
Biological: rAd26-S — Component I (Dose 1) - (0.5 ml per dose) contains:
  Active substance: recombinant adenovirus serotype 26 particles containing the SARS-CoV-2 protein S gene, in the amount of (1.0±0.5) х 10^11 particles per dose (unit dose strength 1 × 10^11 vp/0.5 mL) .
  Solution for intramuscular injection, supplied in vials in containers
  Other Names: Gam-COVID-Vac combined vector vaccine

SUMMARY:
This is a Phase I/II, parallel group, single blinded (participant blinded), randomised study assessing the immunogenicity and safety of AZD1222 and rAd26-S administered as heterologous prime-boost in alternating order in 2 study groups for the Prevention of COVID-19.

DETAILED DESCRIPTION:
This is a prospective, single blinded randomised clinical study, designed to provide data on the heterologous prime boost use of AZD1222 and rAd26-S, to be administered one after the other interchangeably. This study aims to explore the immunogenicity and safety of combining these 2 different adenovirus vector vaccines in the prevention of coronavirus disease 2019 (COVID-19).

Participants will be healthy adults ≥ 18 years of age.

Approximately 100 participants will be randomised (1:1) to one of the following groups:

* Group A: 1 intramuscular (IM) injection of 5×10^10 vp (nominal) of AZD1222 on Day 1 followed by rAd26-S (1.0±0.5) х 10^11vp (nominal) on Day 29.
* Group B: 1 IM injection of rAd26-S (1.0±0.5) х 10^11vp (nominal) on Day 1 followed by AZD1222 5×10^10 vp (nominal) on Day 29.

Immunogenicity will be assessed for the duration of the study, including serologic quantification of severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) antigen specific antibody levels and antibody seroconversion rate, neutralising antibody assays and cellular immunity testing.

Safety will be assessed for the duration of the study as follows:

* Solicited adverse events (AEs) (local and systemic) will be assessed for 7 days following each vaccination (Day 1 through Day 7 for first vaccination and Day 29 through Day 35 for second vaccination).
* Unsolicited AEs will be recorded for 29 days following each vaccination (ie, until Day 29 following the first vaccination and Day 57 following the second vaccination).
* Serious adverse events (SAEs) will be recorded from signing of the informed consent form through Day 180. However, the safety endpoint for SAEs will be assessed after the first vaccination (see Section 12.2).
* Adverse events of special interest (AESIs) will be recorded from first vaccination through Day 180.

This study is going to be conducted in the United Arab Emirates. All participants will remain on study for 6 months (180 days) following the first vaccination.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Participants are:

   * Overtly healthy as determined by medical evaluation, or
   * Medically stable such that, according to the judgment of the investigator, hospitalisation within the study period is not anticipated and the participant appears likely to be able to remain in follow-up through the end of protocol-specified follow up.

   (A stable medical condition is defined as disease not requiring significant change in therapy or hospitalisation for worsening disease during the 3 months prior to enrolment.)
2. Able to understand and comply with study requirements/procedures based on the assessment of the investigator.
3. Female participants

   1. Women of childbearing potential must:

      * Have a negative pregnancy test on the day of screening and on Day 1
      * Use one highly effective form of birth control for at least 28 days prior to Day 1 and agree to continue using one highly effective form of birth control through 60 days following administration of the second dose of study vaccine. A highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly. Periodic abstinence, the rhythm method, and withdrawal are NOT acceptable methods of contraception.
   2. Women are considered of childbearing potential unless they meet either of the following criteria:

      * Surgically sterilised (including bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or
      * Postmenopausal
      * For women aged < 50 years, postmenopausal is defined as having both:

        * A history of ≥ 12 months amenorrhea prior to first dosing, without an alternative cause, following cessation of exogenous sex-hormonal treatment, and
        * A follicle-stimulating hormone level in the post-menopausal range (Until follicle-stimulating hormone is documented to be within menopausal range, the participant is to be considered of childbearing potential.)
      * For women aged ≥ 50 years, postmenopausal is defined as having a history of ≥ 12 months amenorrhea prior to first dosing, without an alternative cause, following cessation of exogenous sex-hormonal treatment.
4. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol of the sudy.

Exclusion Criteria:

1. Known past laboratory-confirmed SARS-CoV-2 infection less than 6 month prior to screening (the date of diagnosis must be confirmed by an official document).
2. Positive severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) reverse transcription-polymerase chain reaction (RT-PCR) test at screening.
3. Significant infection or other illness, including fever > 37.8°C on the day prior to or day of randomisation.
4. Any confirmed or suspected immunosuppressive or immunodeficient state, including human immunodeficiency virus (HIV) infection; asplenia; recurrent severe infections and use of chronic immunosuppressant medication within the past 6 months (≥ 20 mg/day of prednisone or its equivalent, given daily or on alternate days for ≥ 15 days within 30 days prior to vaccination), except topical/inhaled steroids or short term oral steroids (course lasting ≤ 14 days).

   1. Note: HIV-positive participants with CD4 counts > 500 for ≥ 12 months and on a stable HIV antiretroviral regimen may be enrolled.
   2. Note: Topical tacrolimus is allowed if not used within 14 days prior to the day of enrolment.
5. History of allergy to any component of the vaccine.
6. Any history of anaphylaxis or angioedema.
7. Current diagnosis of or treatment for cancer (except basal cell carcinoma of the skin and uterine cervical carcinoma in situ).
8. History of serious psychiatric condition likely to affect participation in the study.
9. Bleeding disorder (eg, factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture.
10. Suspected or known current alcohol or drug dependency.
11. History of Guillain-Barré syndrome or any other demyelinating condition.
12. Any other significant disease, disorder or finding which may significantly increase the risk to the participant because of participation in the study, affect the ability of the participant to participate in the study or impair interpretation of the study data.

    (Note: The adverse events of special interest (AESIs) as outlined in Appendix F of the protocol should be considered when evaluating a participant for Exclusion Criterion 13, as the presence of these AESIs, especially if untreated or uncontrolled, may be a safety risk to the participant, affect the ability of the participant to participate in the study or impair interpretation of the study data. Investigators should review and consider the list of conditions in Appendix F. If any of these conditions is present in a participant, the Investigator is asked to utilise his/her clinical judgment in determining the participant's eligibility for the study. Should the participant have conditions as outlined in Appendix F and is enrolled, the Investigator is asked to document notes on site regarding the final rationale for enrolment.)
13. Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder and neurological illness (mild/moderate well controlled comorbidities are allowed).
14. Prior splenectomy.
15. History of cerebral venous sinus thrombosis or experienced major venous and/or arterial thrombosis.
16. Receipt of any vaccine (licensed or investigational) other than the study vaccine within 30 days before and after each study vaccination.
17. Prior (less than 12 months) or planned receipt of an investigational or licensed vaccine or product likely to impact on interpretation of the trial data (eg, adenovirus vectored vaccines, any coronavirus vaccines).

    (Note: Participant vaccinated against coronavirus 12 months or more prior to screening could be included.)
18. Administration of immunoglobulins and/or any blood products within the 3 months preceding the planned administration of the vaccine candidate.
19. Continuous use of anticoagulants, such as coumarins and related anticoagulants (ie, warfarin) or novel oral anticoagulants (ie, apixaban, rivaroxaban, dabigatran and edoxaban).
20. Participation in COVID-19 prophylactic drug trials for the duration of the study.
21. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca/R-Pharm staff and/or staff at the study site).
22. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
23. Previous randomisation in the present study.
24. For women only - currently pregnant (confirmed with positive pregnancy test) or breast feeding.
25. Unwilling to refrain from blood donation during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Antibody seroconversion rate (≥ 4 fold increase from baseline) against SARS-CoV-2 Spike protein 29 days post second vaccination | Day 57
  The proportion of participants with post treatment seroresponse (defined as ≥ 4-fold rise in titres from Day 1 baseline value) to S antigen 29 days post second vaccination.

SECONDARY OUTCOMES:
Incidence of local and systemic solicited Adverse Events (AEs) for 7 days following each vaccination | from Day 1 till Day 7 and from Day 29 till Day 35
  Number of Participants Reporting local (Pain at the site of injection, Erythema/redness at the site of injection, Tenderness, Induration/swelling at the site of injection) and systemic (Fever > 37.8°C, Chills, Muscle pains, Fatigue, Headache, Malaise, Nausea, Vomiting) Solicited Adverse Events for 7 days following each vaccination (Day 1 through Day 7 for first vaccination and Day 29 through Day 35 for second vaccination)
Incidence of unsolicited AEs, Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) through 29 days post each vaccination | from day 1 till Day 29 and from Day 29 till Day 57
  Number of Participants Reporting unsolicited AEs, SAEs and AESIs through 29 days post each vaccination.
Antibody seroconversion rate (≥ 4 fold increase from baseline) against SARS-CoV-2 Spike protein 29 days post first vaccination | Day 29
  The proportion of participants who have a post treatment seroresponse (defined as: ≥ 4 fold rise in titres from Day 1 baseline value) to the S antigens 29 days post first vaccination.
Antibody seroconversion rate (≥ 4 fold increase from baseline) against Receptor Binding Domain (RBD) antigen | Day 29, Day 57
  The proportion of participants with post treatment seroresponse (defined as: ≥ 4-fold rise in titres from Day 1 baseline value) to RBD antigen 29 days post each vaccination.
Сhange from baseline Geometric Mean Titre (GMT) of immunogenicity against Spike and RBD antigens at Day 15, 29, 57, 180. | Day 1, Day 15, Day 29, Day 57, Day 180
  Сhange from baseline GMT against S and RBD antigens at at Day 15, 29, 57, 180.
Change from baseline Geometric Mean Fold Rise (GMFR) of immunogenicity against Spike and RBD antigens at Day 15, 29, 57, 180. | Day 1, Day 15, Day 29, Day 57, Day 180
  Change from baseline GMFR against S and RBD antigens at Day 15, 29, 57, 180.
Antibody seroconversion rate (≥ 4 fold increase from baseline) SARS-CoV-2 neutralising antibodies 29 days post each vaccination (Day 29 and Day 57) | Day 29, Day 57
  The proportion of participants with post treatment seroresponse (defined as: ≥ 4-fold rise in titres day from Day 1 baseline value to 29 days post each vaccination - Day 29 and Day 57), as measured by SARS-CoV-2 neutralising antibodies
Change from baseline GMT of immunogenicity as measured by SARS-CoV-2 neutralising antibodies at Day 15, 29, 57, 180. | On Day 1, Day 15, Day 29, Day 57, Day 180
  Change from baseline GMT of immunogenicity as measured by SARS-CoV-2 neutralising antibodies at Day 15, 29, 57, 180.
Change from baseline GMFR of immunogenicity as measured by SARS-CoV-2 neutralising antibodies at Day 15, 29, 57, 180. | On Day 1, Day 15, Day 29, Day 57, Day 180
  Change from baseline GMFR of immunogenicity as measured by SARS-CoV-2 neutralising antibodies at Day 15, 29, 57, 180.
Change from baseline the number of proliferating CD4 and CD8 cells in response to mitogen stimulation and their ratio in trial subjects. | Day 1, Day 29, Day 57
  The number of proliferating CD4 and CD8 cells in response to mitogen stimulation and their ratio in trial subjects at Day 1, Day 29 and Day 57.
Change from baseline Interferon gamma concentration in response to S Ag simulation | Day 1, Day 29, Day 57
  Interferon gamma concentration in response to S Ag simulation at Day 1, Day 29 and Day 57.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — Chief Medical Officer, R-Pharm
Locations (1):
- Tawam Hospital, Al Ain City, United Arab Emirates